CLINICAL TRIAL: NCT05599477
Title: The GATE Study: Endoscopic Sutured Gastroplasty in Type 2 Diabetic, Obese Patients
Brief Title: The GATE Study: Endoscopic Sutured Gastroplasty in Type 2 Diabetic, Obese Patients Using the Endomina Device
Acronym: GATE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Endotools Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL82297.091.22
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Diabete Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic sutured gastroplasty (Experimental)
  Interventions: Device: Endoscopic sutured gastroplasty with endomina

INTERVENTIONS:
Device: Endoscopic sutured gastroplasty with endomina — The endomina is is used to perform endoscopic sutured gastroplasty. Two guidewires are introduced via an upper GI endoscopy down to the duodenum. The endomina system is introduced and the endoscope is inserted and fixed to the system. Next a needle preloaded with suture is introduced into the platform. The stomach wall is grasped with a forceps and pulled back. The needle is pushed through the wall, and a first tag is released. The needle is retracted, the first plicature is released and a second plicature is made with the same needle at the opposite wall. Then the pretied knot is grasped and tightened until both plicatures are firmly apposed. The same procedure is repeated along the great curvature from the incisura to the upper body.
  The procedure will include the placement of 6-9 sutures. The first suture is done at the level of the incisura, at the lower part of the greater curvature. The following stitches are placed along the body of the stomach
  Other Names: Endoscopic sleeve gastroplasty

SUMMARY:
Rationale: Diabetes mellitus is a chronic disease that is often associated with long-term macrovascular and microvascular complications and decreased life expectancy. Approximately 70% of patients with type 2 diabetes mellitus (DM2) are overweight or obese. Weight loss benefits several aspects of DM2, such as improved glycemic control, increased insulin sensitivity and reduced fasting insulin. This results in a reduction in glycated hemoglobin. Interventions for weight loss in patients with DM2 include diet, exercise, but also pharmacotherapy and bariatric surgery. Current standard pharmacotherapeutic treatment for patients with DM2 in the Netherlands starts with metformin, followed by insulin. Bariatric surgery is indicated at a BMI > 35 kg/m², in combination with other comorbidities. It is associated with better glycemic control and more weight reduction, compared to intensive medical treatment alone. For patients with not adequately controlled DM2 who are not eligible for surgery (i.e., BMI of < 35 kg/m²), there is currently a therapeutic gap, which could be filled by one of the currently available endoscopic therapies aiming to reduce weight. One of these therapies is endoscopic suture gastroplasty, performed with the endomina device (EndoTools Therapeutics S.A.).

Objective: To evaluate the efficacy and safety of endoscopic sutured gastroplasty with the endomina device (EndoTools Therapeutics S.A.) for glycemic control, in obese patients (BMI of 30-40 kg/m²) with DM2 under insulin therapy with or without hypertension.

Study design: Prospective interventional study Study population: All consecutive patients, with a BMI between 30 and 40 kg/m² with DM2 for less than 10 years, treated with insulin therapy.

Intervention: Endoscopic suture gastroplasty will be performed using the endomina device.

Main study parameters/endpoints: Reduction of 0.7% in HbA1C after 1 year post procedure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will undergo endoscopic suture gastroplasty using endomina, which is known with only minor adverse events (abdominal cramps, nausea, vomiting), and a serious adverse events so far of > 1% (one readmission, no surgical intervention needed, no mortality). Afterwards, patients will be followed at 14 days, 1 month, and 3, 6, 9 and 12 months after gastroplasty for clinical and adverse event assessment. Clinical assessment consists of laboratory tests and the quality-of-life questionnaire (EQ-5D-5L), and Diabetes Treatment Satisfaction Questionnaire as well as Quality adjusted life years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years;
* Diagnosed with DM2

  * since at least 1 year
  * but diagnosed no longer than 10 years ago
  * currently under stable dose of insulin for at least 6 months
* HbA1c level of 7.0-11.0% (53-75 mmol/mol) prior to inclusion
* BMI of 30-40 kg/m² with or without hypertension
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol (including compliance to treatment, dietary follow up, visits as scheduled and all study specific procedures)
* Must be able to understand and be willing to provide written informed consent
* Must be eligible for general anesthesia or deep sedation with propofol

Exclusion Criteria:

* Achalasia and any other esophageal motility disorders
* Severe esophagitis (grade C or D)
* Gastro-duodenal ulcer
* GI stenosis or obstruction
* Any history of esophageal or gastric surgery
* Heart diseases: unstable angina, myocardial infarction within the past year, or heart disease classified within the New York Heart Association's Class III or IV functional capacity
* Uncontrolled hypertension (systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg under medication) during last 3 months;
* Severe renal, hepatic, pulmonary disease or cancer (cancer in the past 5 years, except basal cell carcinoma)
* Pregnancy, breast feeding or desire for pregnancy in the coming 12 months
* Any previous bariatric surgery, or endoscopic obesity-related intervention (including POSE, OverStitch, etc.). Intragastric balloon removed within the last 6 months
* Planned gastric surgery 60 days post intervention
* Anticoagulant therapy that cannot be temporarily stopped at the time of the procedure.
* Currently participating in other study (involving change of treatment) that did not reach its primary endpoint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in HbA1c | 1 year
  a reduction of HbA1C of at least 0.7%

SECONDARY OUTCOMES:
Rate of Serious Adverse Events (SAE) and Serious Adverse Device Effects (SADE) during and post procedure | 1 year
Adverse events up to 1-month follow-up for subjects undergoing the procedure under procedural sedation with propofol | 1 year
Cardiovascular events (stroke/TIA, myocardial infarction, admission for heart failure) and all-cause mortality | 1 year
Reduction of HbA1C at 14 days, 1 month, 3, 6, and 9 months after ESG | 1 year
Reduction in fasting plasma glucose levels at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
Proportion of subjects with reduced number and/or reduced dose(s) of diabetes medication at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
Proportion of subjects with mean % excess weight loss (EWL) of more than 25% at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
Proportion of subjects with mean % total body weight loss (TBWL) of more than 5% at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
Decrease in blood pressure expressed in mmHg at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
EQ-5D-5L at 14 days, 1 month, 3, 6 and 12 months after ESG | 1 year
Diabetes Treatment Satisfaction Questionnaire at 14 days, 1 month, 3, 6, 9 and 12 months after ESG | 1 year
Quality adjusted life years (QALYs) | 1 year
Costs and cost-effectiveness. | 1 year
  Costs including health care recourses used (including intervention including endomina device and TAPES, hospital admissions, visits to specialists and GP, emergency room visits, medications used), costs for insulin therapy (including medication, administration, glycemia measurement material)

IPD SHARING:
Plan to Share IPD: Undecided